CLINICAL TRIAL: NCT01011465
Title: The Biology of Resilience: Oxytocin, Social Relationships and Health
Brief Title: The Biology of Resilience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Laura Kubzansky, Associate Professor, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1R21AG030632-01A2 (NIH)
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Results first posted 2012-11-26 (Estimated); Last update posted 2012-11-26 (Estimated); Status verified 2012-10

CONDITIONS: Oxytocin; Placebo
Keywords: Stress; Oxytocin; Social Support; Resilience
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Oxytocin (Experimental): One primary experimental manipulation is the receipt of intranasal oxytocin vs placebo spray prior to participation in a psychosocial stress protocol
  Interventions: Drug: intranasal oxytocin; Behavioral: Social support; Behavioral: No Social Support
- Placebo (Placebo Comparator): The comparison condition for receipt of oxytocin is receipt of a saline intranasal spray
  Interventions: Drug: Placebo; Behavioral: Social support; Behavioral: No Social Support
- Social Support (Experimental): Participants bring a friend to the laboratory who sits with them while they engage in the stress protocol tasks
  Interventions: Drug: intranasal oxytocin; Drug: Placebo; Behavioral: Social support
- No Social Support (Placebo Comparator): Individuals in this condition do not have a friend present while they are engaging in the laboratory protocol.
  Interventions: Drug: intranasal oxytocin; Drug: Placebo; Behavioral: No Social Support
- Female Gender (Other): Effects of oxytocin and social support are examined among women versus men
  Interventions: Drug: intranasal oxytocin; Drug: Placebo; Behavioral: Social support; Behavioral: No Social Support
- Male Gender (Other): Consider effects of oxytocin and social support in men versus women
  Interventions: Drug: intranasal oxytocin; Drug: Placebo; Behavioral: Social support; Behavioral: No Social Support

INTERVENTIONS:
Drug: intranasal oxytocin — The aqueous form of oxytocin (oxytocin injection, synthetic) in 10 ml vials is inserted into a spray bottle. The spray bottle is calibrated so that emptying the spray bottle results in delivering 24 IU of oxytocin. No dilution of the original aqueous form of the oxytocin is necessary. 24 IU of oxytocin will be administered at one time only during the procedure. Approximately half the dose will be sprayed into each nostril. Administration will stop after 24 IUs of oxytocin have been administered. Duration of administration is anticipated to be 2-5 minutes
  Other Names: Pitocin
  Arms: Female Gender; Male Gender; No Social Support; Oxytocin; Social Support
Drug: Placebo — Participants in the placebo condition receive an equivalent amount of saline for intranasal spray administration. The placebo will be administered at one time only during the procedure. Approximately half the dose will be sprayed into each nostril. Administration will stop after the full amount in the spray bottle has been used. Duration of administration is anticipated to be 2-5 minutes
  Arms: Female Gender; Male Gender; No Social Support; Placebo; Social Support
Behavioral: Social support — Prior to coming to the laboratory, participants are randomly assigned to one of two conditions, requiring them to appear alone or accompanied by a partner. If instructed to bring a same-sex close friend (excluding spouses, participants are joined by their support partners join participants at the start of the stress exposure. The social support condition includes a number of strategies designed to standardize the type of support available to participants across individuals.
  Arms: Female Gender; Male Gender; Oxytocin; Placebo; Social Support
Behavioral: No Social Support — Prior to coming to the laboratory, participants are randomly assigned to one of two conditions, requiring them to appear alone or accompanied by a partner. They are then instructed to bring a same-sex close friend (excluding spouses) with them, or to come alone. If they come to the laboratory without a friend, they engage in all the laboratory procedures without a friend present.
  Arms: Female Gender; Male Gender; No Social Support; Oxytocin; Placebo

SUMMARY:
Positive social relationships have consistently been associated with better health, although the neurobiological underpinnings of these observed effects remain largely unknown. The overall goal of the proposed work is to explore novel biological pathways that may explain how social relationships influence health. Recent theorizing suggests that the oxytocin system may underlie some of the observed beneficial effects. Four hypotheses will be examined:

1. Oxytocin ameliorates the deleterious neuroendocrine, cardiovascular, and subjective effects of stress.
2. Oxytocin and social support have similar and additive stress-buffering effects.
3. Effects of oxytocin are evident among younger and older adults.
4. Effects of oxytocin are stronger in women vs men.

DETAILED DESCRIPTION:
Positive social relationships have consistently been associated with better health, although the neurobiological underpinnings of these observed effects are not well understood. Valuable insight may be gained by a life course perspective as it is becoming increasingly apparent that early life social experiences are crucially related to later life functioning and well-being. The overall goal of the proposed work is to explore novel biological pathways that help to explain how social relationships influence health. Recent theorizing on the biology relating positive social and emotional factors to health and patterns of resilience suggest that the oxytocin system may underlie some of the observed beneficial effects. Historically, most work on the oxytocin system in humans has been tied to reproductive outcomes (e.g., lactation), with more limited work on children and young adults. A growing body of experimental research with animals suggests that early in life, oxytocin not only creates powerful social bonds between a mother and child but may also stimulate growth and restorative processes as well as buffer deleterious stress-related neuroendocrine activation throughout the life course. Moreover, the animal literature has suggested that oxytocin is more potent in the presence of higher estrogen levels, leading investigators to hypothesize that effects of oxytocin are stronger in women than men, but few studies have tested this hypothesis in humans. A better understanding of the inter-relationships between oxytocin, social relationships, stress, and health will be gained by examining these factors in a controlled laboratory setting. The immediate goal of this research is to determine whether oxytocin plays a critical role in determining neuroendocrine, cardiovascular, and subjective responses to stress across age and gender, and to examine the effects of oxytocin in relation to those of social support. To achieve these goals, experimental research is proposed to examine the effects of exogenously administered (intranasal) oxytocin on psychological and physiological outcomes, under conditions of stress. The specific aims of this exploratory project are to test the following hypotheses:

1. Oxytocin ameliorates the deleterious neuroendocrine, cardiovascular, and subjective effects of stress.
2. Oxytocin and social support have similar and additive stress-buffering effects.
3. Effects of oxytocin are stronger in women versus men.
4. Effects of oxytocin are similar across a range of younger and older adult ages.

Hypotheses will be tested via a placebo-controlled double blind study using a sample of healthy men and women recruited from the community (overall n = 320). The proposed experimental study will consider oxytocin effects on a range of outcomes. These include autonomic reactivity as measured by blood pressure responses and high frequency heart rate variability (measure of vagal tone). Stress-related cardiovascular phenotypes as characterized by the patterning of ventricle contractility, vascular resistance, and cardiac output will also be assessed. Other outcomes include measures of neuroendocrine effects as measured by levels of cortisol and dehydroepiandrosterone (DHEA) hormone, subjective distress and positive affect. Participants will be randomly assigned to receive either exogenous oxytocin or placebo. They will undergo a social stress manipulation with or without social support (randomly assigned), and outcome measures will be obtained at multiple times during the experimental procedure. The experiment will test whether effects of oxytocin and social support are similar and additive, and will also compare effects of oxytocin and social support across men and women of varying ages. This multidisciplinary study uses a biobehavioral framework to examine interactions between psychological, social, and biological levels of functioning, and is informed by theories of how key early life exposures may impact health over the life course. The provision of an R21 award for this work will facilitate novel research that could have a major impact on our understanding of whether and how oxytocin influences responses to stress in humans. The proposed exploratory research will lay the groundwork for the submission of an R01 grant proposal that will have greater resources for addressing both the questions that cannot be addressed with this more limited mechanism as well as new questions that will undoubtedly arise. Ultimately we expect this project will provide a solid platform from which to launch a larger program of research aimed at identifying how positive social and emotional experiences influence adult health and longevity. A neurobiological understanding of resilience can inform efforts for both prevention and intervention of diseases or problems common in later life.

ELIGIBILITY:
Inclusion Criteria:

* age 22-65, BMI < 30, healthy, English-speaking, 9th grade reading level.

Exclusion Criteria:

* any known medical condition (including mental disorders) or on any type of medication
* high levels of social anxiety
* smokers
* high rates of alcohol or drug use
* pregnant or suspected pregnant
* breastfeeding
* blood pressures > 140/90 mm Hg
* subject does not have a close friend available to participate in the study with him/her

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2009-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura D Kubzansky, PhD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Harvard School of Public Health, Boston, Massachusetts, United States

REFERENCES:
- [Background] Kubzansky LD, Mendes WB, Appleton A, Block J, Adler GK. Protocol for an experimental investigation of the roles of oxytocin and social support in neuroendocrine, cardiovascular, and subjective responses to stress across age and gender. BMC Public Health. 2009 Dec 21;9:481. doi: 10.1186/1471-2458-9-481. PMID 20025778
- [Result] Kubzansky LD, Mendes WB, Appleton AA, Block J, Adler GK. A heartfelt response: Oxytocin effects on response to social stress in men and women. Biol Psychol. 2012 Apr;90(1):1-9. doi: 10.1016/j.biopsycho.2012.02.010. Epub 2012 Feb 23. PMID 22387929

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in this study from 6/2008 to 4/2012. Initial screening was done by phone and email. Medical screening took place at a hospital clinic and the rest of the study took place at the Harvard School of Public Health.
Pre-assignment Details: After initial screening , participants were asked to sign consent form and screened in a medical clinic prior to group assignment. Participants were excluded for violating study criteria, including having BMI>30, high blood pressure, acute illness, smoking or drug use and chronic medical conditions. Refusal to sign consent also led to exclusion.
Groups:
- Female, OT, Alone: Effects of intranasal oxytocin and social support examined among women versus men.
  Intranasal oxytocin : The aqueous form of oxytocin (oxytocin injection, synthetic) in 10 ml vials is inserted into a spray bottle. The spray bottle is calibrated so that emptying the spray bottle results in delivering 24 IU of oxytocin. No dilution of the original aqueous form of the oxytocin is necessary. 24 IU of oxytocin is administered.
  Social support - Alone : Prior to lab visit, participant is randomly assigned to one of two conditions, requiring them to appear alone or accompanied by partner. Participant assigned to alone is unaccompanied during tasks.
- Female, OT, Friend: Effects of intranasal oxytocin and social support examined among women versus men.
  Intranasal oxytocin : The aqueous form of oxytocin (oxytocin injection, synthetic) in 10 ml vials is inserted into a spray bottle. The spray bottle is calibrated so that emptying the spray bottle results in delivering 24 IU of oxytocin. No dilution of the original aqueous form of the oxytocin is necessary. 24 IU of oxytocin is administered.
  Social support - Friend : Prior to lab visit, participant is randomly assigned to one of two conditions, requiring them to appear alone or accompanied by partner. If instructed to bring a same-sex close friend (excluding spouses), participants are joined by their support partners at the start of the stress exposure. The social support condition includes a number of strategies designed to standardize the type of support available to participants across individuals.
- Female, Placebo, Alone: Effects of intranasal oxytocin and social support examined among women versus men.
  Placebo : Participants in the placebo condition receive an equivalent amount of saline for intranasal spray administration. The placebo is administered at one time only during the procedure. Approximately half the dose is sprayed into each nostril. Administration stops after the full amount in the spray bottle has been used.
  Social support - Alone : Prior to lab visit, participant is randomly assigned to one of two conditions, requiring them to appear alone or accompanied by partner. Participant assigned to alone is unaccompanied during tasks.
- Female, Placebo, Friend: Effects of intranasal oxytocin and social support examined among women versus men.
  Placebo : Participants in the placebo condition receive an equivalent amount of saline for intranasal spray administration. The placebo is administered at one time only during the procedure. Approximately half the dose is sprayed into each nostril. Administration stops after the full amount in the spray bottle has been used.
  Social support - Friend : Prior to lab visit, participant is randomly assigned to one of two conditions, requiring them to appear alone or accompanied by partner. If instructed to bring a same-sex close friend (excluding spouses), participants are joined by their support partners at the start of the stress exposure. The social support condition includes a number of strategies designed to standardize the type of support available to participants across individuals.
- Male, OT, Alone: Effects of intranasal oxytocin and social support examined among men versus women.
  Intranasal oxytocin : The aqueous form of oxytocin (oxytocin injection, synthetic) in 10 ml vials is inserted into a spray bottle. The spray bottle is calibrated so that emptying the spray bottle results in delivering 24 IU of oxytocin. No dilution of the original aqueous form of the oxytocin is necessary. 24 IU of oxytocin is administered.
  Social support - Alone : Prior to lab visit, participant is randomly assigned to one of two conditions, requiring them to appear alone or accompanied by partner. Participant assigned to alone is unaccompanied during tasks.
- Male, OT, Friend: Effects of intranasal oxytocin and social support examined among men versus women.
  Intranasal oxytocin : The aqueous form of oxytocin (oxytocin injection, synthetic) in 10 ml vials is inserted into a spray bottle. The spray bottle is calibrated so that emptying the spray bottle results in delivering 24 IU of oxytocin. No dilution of the original aqueous form of the oxytocin is necessary. 24 IU of oxytocin is administered.
  Social support - Friend : Prior to lab visit, participant is randomly assigned to one of two conditions, requiring them to appear alone or accompanied by partner. If instructed to bring a same-sex close friend (excluding spouses), participants are joined by their support partners at the start of the stress exposure. The social support condition includes a number of strategies designed to standardize the type of support available to participants across individuals.
- Male, Placebo, Alone: Effects of intranasal oxytocin and social support examined among men versus women.
  Placebo : Participants in the placebo condition receive an equivalent amount of saline for intranasal spray administration. The placebo is administered at one time only during the procedure. Approximately half the dose is sprayed into each nostril. Administration stops after the full amount in the spray bottle has been used.
  Social support - Alone : Prior to lab visit, participant is randomly assigned to one of two conditions, requiring them to appear alone or accompanied by partner. Participant assigned to alone is unaccompanied during tasks.
- Male, Placebo, Friend: Effects of intranasal oxytocin and social support examined among men versus women.
  Placebo : Participants in the placebo condition receive an equivalent amount of saline for intranasal spray administration. The placebo is administered at one time only during the procedure. Approximately half the dose is sprayed into each nostril. Administration stops after the full amount in the spray bottle has been used.
  Social support - Friend : Prior to lab visit, participant is randomly assigned to one of two conditions, requiring them to appear alone or accompanied by partner. If instructed to bring a same-sex close friend (excluding spouses), participants are joined by their support partners at the start of the stress exposure. The social support condition includes a number of strategies designed to standardize the type of support available to participants across individuals.
Period: Overall Study
Arm/Group | Female, OT, Alone | Female, OT, Friend | Female, Placebo, Alone | Female, Placebo, Friend | Male, OT, Alone | Male, OT, Friend | Male, Placebo, Alone | Male, Placebo, Friend
Started | 36 | 20 | 36 | 18 | 47 | 29 | 52 | 32
Completed | 34 | 19 | 36 | 18 | 46 | 29 | 51 | 32
Not Completed | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Female, OT, Alone | Female, OT, Friend | Female, Placebo, Alone | Female, Placebo, Friend | Male, OT, Alone | Male, OT, Friend | Male, Placebo, Alone | Male, Placebo, Friend | Total
Number analyzed (Participants) | 36 | 20 | 36 | 18 | 47 | 29 | 52 | 32 | 270
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 36 | 20 | 36 | 18 | 47 | 29 | 52 | 32 | 270
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.9 (11.2) | 28.7 (6.2) | 34.3 (10.7) | 33.7 (13.2) | 34.8 (11.8) | 28.4 (9.0) | 36.0 (12.1) | 32.4 (9.7) | 33.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 20 | 36 | 18 | 0 | 0 | 0 | 0 | 110
  Male | 0 | 0 | 0 | 0 | 47 | 29 | 52 | 32 | 160
Region of Enrollment [Number; unit: participants]
  United States | 36 | 20 | 36 | 18 | 47 | 29 | 52 | 32 | 270

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure Change From Baseline to Second Stress Task Experience - Autonomic Stress Response Measure
Description: Systolic blood pressure (SBP)is connected with reaction to exposure to stress. Systolic blood pressure is collected at baseline and after nasal spray administration/directly before stress tasks; it represents anticipatory stress reaction. This measure represents the difference between baseline and pre-task systolic blood pressure values. A greater difference score represents an increase from baseline in systolic blood pressure during the pre-task, and so a larger difference score represents higher reactivity. A lower difference score, or negative difference score, indicates a lower increase, or even decrease, from baseline in systolic blood pressure during the pre-task and reflects less reactivity. Reactivity is associated with increased risk of developing hypertension. Range of baseline/pre-count differences in SBP: -11 to 37.7
Time Frame: within 2 hours of treatment
Population: All participants who received oxytocin or placebo, who completed the study, had relevant covariate data, and for whom systolic blood pressure was collected, were included
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Oxytocin Group: Intranasal oxytocin : The aqueous form of oxytocin (oxytocin injection, synthetic) in 10 ml vials is inserted into a spray bottle. The spray bottle is calibrated so that emptying the spray bottle results in delivering 24 IU of oxytocin. No dilution of the original aqueous form of the oxytocin is necessary. 24 IU of oxytocin is administered.
- Placebo Group: Placebo : Participants in the placebo condition receive an equivalent amount of saline for intranasal spray administration. The placebo is administered at one time only during the procedure. Approximately half the dose is sprayed into each nostril. Administration stops after the full amount in the spray bottle has been used.
- Female: Effects of stress exposure examined among women versus men
- Male: Effects of stress exposure examined among men versus women
- Social Support - Alone: Social support - Alone : Prior to lab visit, participant is randomly assigned to one of two conditions, requiring them to appear alone or accompanied by partner. Participant assigned to alone is unaccompanied during tasks.
- Social Support - Friend: Social support - Friend : Prior to lab visit, participant is randomly assigned to one of two conditions, requiring them to appear alone or accompanied by partner. If instructed to bring a same-sex close friend (excluding spouses), participants are joined by their support partners at the start of the stress exposure. The social support condition includes a number of strategies designed to standardize the type of support available to participants across individuals.
Arm/Group | Oxytocin Group | Placebo Group | Female | Male | Social Support - Alone | Social Support - Friend
Number analyzed (Participants) | 54 | 55 | 43 | 66 | 61 | 48
mm Hg | 9.4 (8.2) | 12.9 (7.9) | 11.3 (9.3) | 11.1 (7.5) | 10.7 (7.4) | 11.7 (9.2)
Statistical Analysis 1: Comparison: Oxytocin Group vs Placebo Group; The null hypothesis is that both groups will have similar rise in SBP in response to stress; Test type: Superiority or Other; p = 0.03, t-test, 2 sided; Mean Difference (Final Values) = 3.4
Statistical Analysis 2: Comparison: Female vs Male; The null hypothesis is that both groups will have similar rise in SBP in response to stress; Test type: Superiority or Other; p = 0.89, t-test, 2 sided; Mean Difference (Final Values) = -0.23
Statistical Analysis 3: Comparison: Social Support - Alone vs Social Support - Friend; The null hypothesis is that both groups will have similar rise in SBP in response to stress; Test type: Superiority or Other; p = 0.52, t-test, 2 sided; Mean Difference (Final Values) = -1.01

2. Primary Outcome: Difference of Pre-count and Baseline Self-reported Negative Affect (Using Negative Sub-scale of Positive and Negative Affect Schedule (PANAS) Measure).
Description: Based on 20-item Positive and Negative Affect Schedule (PANAS) which comprises two mood scales, positive affect and negative affect. Each item is rated on a 5-point scale ranging from (1 = very slightly or not at all) to (5 = extremely) to indicate how the respondent felt at the moment the question was asked. Here, we've used the negative affect sub-scale which consists of the sum of the 10 negative affect items, with a possible range of 10 (least negative affect) to 50 (most negative affect). This score was measured at baseline (study range: 10 to 29) and directly before stress exposure (study range: 10 to 37), and the reported value is the difference between these two scores (range of differences: -13 to 26). It estimates negative affect due to anticipatory stress. The value is the difference between the pre-stress measure and baseline measure, therefore a larger number for the difference means a bigger increase in negative affect due to anticipatory stress, and is a worse outcome.
Time Frame: 2 hours
Population: All participants who received oxytocin or placebo, who completed the study, had relevant covariate data, and for whom negative affect score was calculated, were included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin Group | Placebo Group | Female | Male | Social Support - Alone | Social Support - Friend
Number analyzed (Participants) | 125 | 129 | 102 | 152 | 158 | 96
units on a scale | 1.4 (4.5) | 1.8 (4.1) | 2.1 (4.7) | 1.2 (3.9) | 1.8 (4.9) | 1.2 (3.1)
Statistical Analysis 1: Comparison: Oxytocin Group vs Placebo Group; The null hypothesis states that both groups will have similar PANAS negative affect score change in response to stress; Test type: Superiority or Other; p = 0.43, t-test, 2 sided; Mean Difference (Final Values) = 0.42
Statistical Analysis 2: Comparison: Female vs Male; The null hypothesis states that both groups will have similar PANAS negative affect score change in response to stress; Test type: Superiority or Other; p = 0.08, t-test, 2 sided; Mean Difference (Final Values) = -0.96
Statistical Analysis 3: Comparison: Social Support - Alone vs Social Support - Friend; The null hypothesis states that both groups will have similar PANAS negative affect score change in response to stress; Test type: Superiority or Other; p = 0.25, ANOVA; Mean Difference (Final Values) = 0.64

3. Primary Outcome: Speech Threat and Challenge
Description: Measure of threat and challenge calculated from observation of non-verbal behavioral cues during stress exposure. Threat (negative reaction) results when an individual does not feel that he or she has sufficient resources to complete a task or manage a difficult situation. Its reverse, challenge (positive reaction), occurs when an individual perceives that he or she has sufficient resources. Independent observers used videotapes of behavior during the stress tasks and rated participants on 7 point scales for 11 challenge-related behaviors (comfortable, confident, enthusiastic, clear, alert, high level of eye contact, etc), and for 8 threat-related behaviors (agitation, rigid posture, speech disfluency, etc). Challenge scores were averaged, and threat scores averaged then reverse-scored. The mean of challenge and reversed threat scores comprise the score used here. Range: 1.1 to 6.1, with higher scores representing more challenge orientation and reflecting a better outcome.
Time Frame: 2 hours
Population: All participants who received oxytocin or placebo, who completed the study, had relevant covariate data, and for whom speech threat score was calculated, were included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin Group | Placebo Group | Female | Male | Social Support - Alone | Social Support - Friend
Number analyzed (Participants) | 111 | 116 | 97 | 130 | 140 | 87
units on a scale | 4.6 (1.0) | 4.6 (1.0) | 4.5 (1.0) | 4.6 (1.0) | 4.6 (0.9) | 4.6 (1.1)
Statistical Analysis 1: Comparison: Oxytocin Group vs Placebo Group; The null hypothesis states that both groups had similar threat/challenge scores during the speech task; Test type: Superiority or Other; p = 0.83, t-test, 2 sided; Mean Difference (Final Values) = -0.03
Statistical Analysis 2: Comparison: Female vs Male; The null hypothesis states that both groups had similar threat/challenge scores during the speech task; Test type: Superiority or Other; p = 0.56, t-test, 2 sided; Mean Difference (Final Values) = 0.08
Statistical Analysis 3: Comparison: Social Support - Alone vs Social Support - Friend; The null hypothesis states that both groups had similar threat/challenge scores during the speech task; Test type: Superiority or Other; p = 0.95, t-test, 2 sided; Mean Difference (Final Values) = 0.01

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study, ~ 3 years
Arm/Group | Female, OT, Alone | Female, OT, Friend | Female, Placebo, Alone | Female, Placebo, Friend | Male, OT, Alone | Male, OT, Friend | Male, Placebo, Alone | Male, Placebo, Friend
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/20 | 0/36 | 0/18 | 0/47 | 0/29 | 0/52 | 0/32
Other Adverse Events (participants affected / at risk) | 0/36 | 0/20 | 0/36 | 0/18 | 0/47 | 0/29 | 0/52 | 0/32

LIMITATIONS AND CAVEATS:
Data collected earlier in the study is missing blood pressure data due to technical problems.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No